CLINICAL TRIAL: NCT04465253
Title: The Use of the Remotivation Process in an Occupational Therapy Program for Breast Cancer-Related Lymphedema: A Feasibility Study
Brief Title: Remotivation Process for Improving Adherence to Lymphedema Treatment Programs in Patients With Breast Cancer-Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18549; NCI-2020-03475 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18549 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Breast Carcinoma; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Practice Guidelines as Topic; Standard of Care; Motivational Interviewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health services research (discussion, interview) (Experimental): Patients participate in a discussion with an occupational therapist via videoconferencing over 15 minutes QW for 4 weeks about their experience with lymphedema and the occupational services they received. After 4 weeks, some patients may also participate in an interview with an occupational therapist via videoconferencing over 60 minutes. During the first week of the study, patients also receive occupational therapy per standard of care.
  Interventions: Other: Best Practice; Behavioral: Motivational Interviewing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo standard of care occupational therapy
  Other Names: standard of care; standard therapy
Behavioral: Motivational Interviewing — Participate in discussions via videoconferencing
  Other Names: MI; Motivational Interviewing Intervention
Behavioral: Motivational Interviewing — Participate in interview via videoconferencing
  Other Names: MI; Motivational Interviewing Intervention
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well the Remotivation Process in an occupational therapy program works in improving adherence to lymphedema treatment programs in patients with breast cancer-related lymphedema. Lymphedema treatment programs are well developed and effective, but adherence to these programs are an issue. The Remotivation Process is a series of techniques that helps guide discussions between occupational therapists and their patients based on their level of motivation. This study uses the Remotivation Process by gathering patients' thoughts about their experience with lymphedema and occupational therapy services to determine their motivation and learn about the barriers they face in order to improve adherence to these programs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. How does remotivation process change daily performance of the lymphedema management techniques? (Quantitative Study) II. How does the Remotivation Process affect the client's manifestation of breast cancer-related lymphedema (BCRL)? (Quantitative Study) III. How does the Remotivation Process affect the client's occupational participation and quality of life? (Quantitative Study) IV. What are the perspectives of patients with BCRL about the self-management program after participating in an occupational therapy using the Remotivation Process? (Qualitative Study) V. What are the perspectives of patients with BCRL about their arm after the occupational therapy program? (Qualitative Study) VI. How do patients with BCRL describe their daily life after occupational therapy? (Qualitative Study)

OUTLINE:

Patients participate in a discussion with an occupational therapist via videoconferencing over 15 minutes once weekly (QW) for 4 weeks about their experience with lymphedema and the occupational services they received. After 4 weeks, some patients may also participate in an interview with an occupational therapist via videoconferencing over 60 minutes. During the first week of the study, patients also receive occupational therapy per standard of care.

After completion of study, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral upper extremity lymphedema following procedures to address breast cancer, able to communicate in English and participate in discussion sessions and follow up for the duration of the study of eight weeks
* Women will be able to participate in work, household responsibilities, and possible child-rearing responsibilities. These are necessary components of quality of life and occupation, which are the primary concepts of interest of the study. The study will include women with varied levels of functional performance status and life expectancy as long as they are willing to participate in a 15-minute discussion once a week in addition to their scheduled occupational therapy sessions at City of Hope (COH)
* The effects of Remotivation Process on the developing fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* The participant should also be receiving occupational therapy services at COH for BCRL during the first week of the study. The participant can be an on-going patient receiving customary occupational therapy services, or a new patient who will be seen for occupational therapy initial evaluation. The study will include patients with BCRL regardless of any other medical treatment they are receiving in addition to occupational therapy. Some participants may only need less than 4 weeks of customary occupational therapy in order to meet their intervention goals. In this case, the participant will still be asked to return at the end of the fourth week for follow up. Data obtained from the outcome measures will be included in quantitative analysis. The participant will also be included in the list of names that will be randomly selected for the 60-minute interview

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection such as cellulitis
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Change in daily performance of the lymphedema management techniques | Baseline up to 4 weeks
  Will be assessed by frequency count that records the number of times the participant performed the self-management program during the first and fourth week of the study, which is a 7-day period.
Change in arm girth measurement | Baseline up to 4 weeks
  Repeated measures analysis of variance will be used to establish significance and compare the pre-test and post-test girth of the affected arm as well as compare the difference between the affected and non-affected arm at pre-test and post-test. Non-parametric tests will be used should the study not meet the assumptions of parametric test. For non-parametric tests in this case, Friedman's analysis of variance will be used to compare girth.
Change in the number of times each patient performed the self-management program | Baseline up to 4 weeks
  Will be compared by a paired t-test.

SECONDARY OUTCOMES:
Change in quality of life | Baseline up to 4 weeks
  Will be measured by the Lymphedema Quality of Life Inventory. Will be compared using paired t-test. Pearson correlation will be used to determine the correlation between the score from the Model of Human Occupation Screening Tool and scores from the Lymphedema Quality of Life Inventory. Non-parametric tests will be used should the study not meet the assumptions of parametric test. For non-parametric tests in this case, Wilcoxon signed-ranks test will be used to compare the pre-test and post test scores. The Spearman's ranks tests will be used to determine the correlation between the score from the Model of Human Occupation Screening Tool and scores from the Lymphedema Quality of Life Inventory. The qualitative phase follows a descriptive phenomenological design. Thematic analysis will be used to analyze data.
Change in occupational performance | Baseline up to 4 weeks
  Will be measured by the Model of Human Occupation Screening Tool. Will be compared using paired t-test. Pearson correlation will be used to determine the correlation between the score from the Model of Human Occupation Screening Tool and scores from the Lymphedema Quality of Life Inventory. Non-parametric tests will be used should the study not meet the assumptions of parametric test. For non-parametric tests in this case, Wilcoxon signed-ranks test will be used to compare the pre-test and post test scores. The Spearman's ranks tests will be used to determine the correlation between the score from the Model of Human Occupation Screening Tool and scores from the Lymphedema Quality of Life Inventory. The qualitative phase follows a descriptive phenomenological design. Thematic analysis will be used to analyze data.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Hite, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States